CLINICAL TRIAL: NCT01014767
Title: CPT-SIOP-2009: Intercontinental Multidisciplinary Registry and Treatment Optimization Study for Patients With Choroid Plexus Tumors
Brief Title: Intercontinental Multidisciplinary Registry and Treatment Optimization Study for Choroid Plexus Tumors
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI departure from coordinating institution
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPT-SIOP-2009
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Brain Cancer; Choroid Plexus Tumors
Keywords: Choroid Plexus Tumors; Brain Tumor; Chemotherapy; Etoposide; Carboplatin; Vincristine; Cyclophosphamide; Methotrexate; Doxorubicin; Cisplatin; Dactinomycin; temozolomide; irinotecan; Pediatrics
MeSH Terms: conditions — Brain Neoplasms; Choroid Plexus Neoplasms | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Dactinomycin; Doxorubicin; Etoposide; Irinotecan; Leucovorin; Methotrexate; Temozolomide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Standard Arm (1) (Experimental): Alternating chemotherapy cycles with etoposide 100 mg/m2 over 1 hour on days 1-5, carboplatin 350 mg/m2 over 2 hours on day 2 and 3, vincristine 1.5 mg/m2 on day 5 alternating with: etoposide 100 mg/m2 over 1 hour on days 1-5, cyclophosphamide 1 g/m2 over 1 hour on day 2 and 3, vincristine 1.5 mg/m2 on day 5. Six blocks are given in 4 week intervals (day1 to day1). Radiation is given between the second and the third cycle only to a small subgroup of patients defined by age histology staging and response to the first to cycles of chemotherapy.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Vincristine
- Doxorubicin/cisplatin arm (2) (Experimental): Doxorubicin 25 mg/m²/day over 12 hrs on days 1-3, Dactinomycin 45 µg/kg/day (max. 2 mg), i.v. on day 1, and Cisplatin 70 mg/m²/d over 6 hrs on day 4, and Vincristine 1.5 mg/m²/day (max. 2 mg), i.v. on days 8, 15. An identical second cycle is started on day 28 if the side effects allow it. The further treatment is identical to the standard arm with four more cycles of chemotherapy following radiation in some of the patients in all treatment arms.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Vincristine
- Methotrexate Arm (3) (Experimental): Methotrexate 5g/m^2 over 24 hours with leucovorin rescue at hour 42 given three times on days 1 15 and 29. The further treatment is identical in all four treatment arms.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Leucovorin; Drug: Methotrexate; Drug: Vincristine
- Temozolomide Irinotecan arm (4) (Experimental): Temozolomide is given at 150 mg/m2/day x 5 days orally and combined with irinotecan 50 mg/m2/day x 5 days as one hour infusions. Two of these cycles are followed by the common radiation - four cycle chemotherapy protocol.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Irinotecan; Drug: Temozolomide; Drug: Vincristine

INTERVENTIONS:
Drug: Carboplatin — Standard Arm, Cycle 2: 350 mg/m2 IV over 2 hours on day 2 and 3
  All Arms, Cycles 4 & 6: 350 mg/m2 IV over 2 hours on day 2 and 3
  Other Names: Paraplatin
Drug: Cisplatin — Cycles 1 & 2: 70 mg/m²/d IV over 6 hours on day 4
  Other Names: Platinol-AQ; Platinol; CDDP
  Arms: Doxorubicin/cisplatin arm (2)
Drug: Cyclophosphamide — Standard Arm, Cycle 1: 1 g/m^2 IV over 1 hour on day 2 and 3
  All Arms, Cycles 3 & 5: 1 g/m^2 IV over 1 hour on day 2 and 3
  Other Names: Cytoxan; Neosar
Drug: Dactinomycin — Cycles 1 & 2: 45 µg/kg/day (max. 2 mg), IV on day 1
  Other Names: Cosmegen; Actinomycin D
  Arms: Doxorubicin/cisplatin arm (2)
Drug: Doxorubicin — Cycles 1 & 2: 25 mg/m²/day IV over 12 hrs on days 1-3
  Other Names: Adriamycin; Rubex
  Arms: Doxorubicin/cisplatin arm (2)
Drug: Etoposide — Standard Arm (1), Cycles 1 & 2:
  100 mg/m2 IV over 1 hour on days 1-5
  All Arms, Cycles 4-6:
  100 mg/m2 IV over 1 hour on days 1-5
  Other Names: VePsid; VP16
Drug: Irinotecan — Temozolomide Irinotecan arm (4), Cycles 1 & 2:
  50 mg/m2/day x 5 days as 1 hour IV infusions
  Other Names: CPT-11; Camptosar
  Arms: Temozolomide Irinotecan arm (4)
Drug: Leucovorin — Given with Methotrexate as leucovorin rescue at hour 42 given three times on days 1, 15 and 29.
  Other Names: Citrovorum; Wellcovin
  Arms: Methotrexate Arm (3)
Drug: Methotrexate — 5g/m2 IV over 24 hours with leucovorin rescue at hour 42 given three times on days 1, 15 and 29.
  Arms: Methotrexate Arm (3)
Drug: Temozolomide — 150 mg/m2/day x 5 days orally and combined with irinotecan 50 mg/m2/day IV x 5 days as one hour infusions.
  Other Names: Temodar
  Arms: Temozolomide Irinotecan arm (4)
Drug: Vincristine — Standard Arm (1), Cycles 1 & 2 : 1.5 mg/m^2 IV over 15 minutes on day 5
  Doxorubicin/cisplatin arm (2), Cycles 1 & 2: 1.5 mg/m^2/day (max. 2 mg), i.v. on days 8, 15
  For all Groups, Cycles 3 - 6: 1.5 mg/m2 IV over 15 minutes on day 5

SUMMARY:
This is a "tissue banking and data review" research study that also has a "clinical" research part:

* The goal of the tissue banking part of this study is to store tissue in a research tissue bank by the International Society for Pediatric Oncology (SIOP) at an international reference center for choroid plexus tumors. The tissue will be used in future research related to cancer.
* The goal of the data review part of this study is to collect information from the medical records of patients with choroid plexus tumors, and to store the information in SIOP databases for use in future research related to cancer.
* The goal of this clinical research study is to compare 4 chemotherapy treatments for choroid plexus tumors. The safety and level of effectiveness of these study treatments will be compared and studied. The study drugs include different combinations of etoposide, carboplatin, vincristine, cyclophosphamide, methotrexate, doxorubicin, cisplatin, dactinomycin, temozolomide, and irinotecan.

DETAILED DESCRIPTION:
Tissue Banking:

If you agree, samples of your leftover tissue (left over from standard care procedures) will be stored in a research tissue bank by SIOP for use in future research related to cancer.

Data Collection:

If you agree, data from your medical record will be sent to SIOP. The data will be stored in secure research databases by SIOP for use in future research related to cancer. One planned use of the databases is to learn how many patients have choroid plexus tumors, what type of choroid plexus tumors patients have, and the results of treatment for different types of choroid plexus tumors.

Other Information:

Before your tissue and/or data is sent to SIOP for storage, your name and any personal identifying information will be coded to protect your privacy. SIOP will not have access to the codes that link the data to your identity. Tufts Medical CEnter will not have oversight of any leftover tissue and/or data that will be stored by SIOP for additional research.

Length of Study:

You will be on-study for as long as you agree to continue having your tissue and/or data used for research.

This is an investigational study. Up to 190 patients will take part in this study. Up to 6 will be enrolled at M. D. Anderson.

Clinical Research:

The Study Drugs:

The study drugs are all designed to interfere with the growth of cancer cells by blocking cell division, which may cause the cells to die.

Radiation Therapy:

Participants who are eligible may also receive radiation therapy during the study. The type of therapy will be "craniospinal" radiation (radiation to the brain and spinal cord) or "focal" radiation (radiation focused on the tumor only). This will be the doctor's decision, and the radiation doctor will discuss this treatment option with you if you are possibly eligible.

Surgery:

Participants who are eligible may also have surgery during the study. This will be if you have tumor remaining after therapy at certain times in the study, and only if the tumor can be surgically removed. This will be the doctor's decision, and the study doctor will discuss this treatment option with you if you are possibly eligible.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to a study group.

This study is being done in 2 phases. If you are one of the first participants to join the study, you will be enrolled in Phase I. There are 4 study groups in Phase I, and you will have an equal chance of being assigned to any of the 4 groups.

If you are one of the later participants to join the study, you will be enrolled in Phase II. There will be 2 study groups in Phase II, and you will have an equal chance of being assigned to either group.

* One of the study groups in Phase II will receive the study drugs that are called "Group 1" below. (Although none of the study drugs are FDA-approved, Group 1's study drugs are considered the standard treatment for choroid plexus tumors.)
* The other study group in Phase II will be the study group from Phase I that had the best results (Group 2, 3, or 4 as described below).

The study drugs in Cycles 1 and 2 are different in all 4 study groups. All 4 study groups receive the same study drugs in Cycles 3-6.

Cycles in this study are 28 days long.

Study Drug Administration:

Group 1:

* In Cycle 1, you will receive cyclophosphamide by vein over 2 hours on Days 2 and 3, etoposide by vein over 1 hour on Days 1-5, and vincristine by vein over 15 minutes on Day 5.
* In Cycle 2, Group 1 will receive etoposide by vein over 1 hour on Days 1-5, carboplatin by vein over 2 hours on Days 2 and 3, and vincristine by vein over 15 minutes on Day 5.

Group 2:

In Cycles 1 and 2, Group 2 will receive doxorubicin by vein over 12 hours on Days 1-3, dactinomycin by vein over 1 hour on Day 1, cisplatin by vein over 6 hours on Day 4, and vincristine over 15 minutes on Days 8 and 15.

Group 3:

Group 3 will receive methotrexate by vein over 24 hours on Days 1 and 15 of Cycle 1 and Day 1 of Cycle 2.

Group 4:

In Cycles 1 and 2, Group 4 will take temozolomide by mouth once a day on Days 1-5 and receive irinotecan by vein over 1 hour on Days 1-5.

All Groups:

* In Cycles 3 and 5, you will receive cyclophosphamide by vein over 2 hours on Days 2 and 3, etoposide by vein over 1 hour on Days 1-5, and vincristine by vein over 15 minutes on Day 5.
* In Cycles 4 and 6, you will receive etoposide by vein over 1 hour on Days 1-5, carboplatin by vein over 2 hours on Days 2 and 3, and vincristine by vein over 15 minutes on Day 5.
* Depending on your and the doctor's decision, the drugs that you receive by vein may be given into a central venous catheter. This is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will sign a separate consent form for it.

Possible Additional Therapies:

Depending on your age and the disease status, you may receive radiation therapy before Cycle 3. The radiation treatments will be once a day, a few minutes each, 5 days a week for about 6 weeks.

If you have tumor remaining after Cycle 1, after radiation therapy, and/or after your last study drug dose, you may have surgery if the tumor can be surgically removed. Your doctor will explain the surgery to you in more detail, and you will sign a separate consent form for it.

Possible Different Type of Etoposide Administration:

If the tumor is in your cerebrospinal fluid (fluid in your brain and spine) and you have not received craniospinal radiation, you will receive etoposide "intrathecally" rather than by vein. This means the drug will be given directly into your cerebrospinal fluid. This will be done on Days 1 and 28 of every cycle. Your doctor will explain the intrathecal injection procedure to you in more detail, and you will sign a separate consent form for it.

In this case, etoposide may (depending on your and the doctor's decision) be given into an Ommaya reservoir or Rickham capsule. These are devices that are surgically placed under the scalp so that the drug can be given directly into your cerebrospinal fluid. If this applies to you, the surgeon will explain the surgery to you in more detail, and you will sign a separate consent form for it.

Drugs to Prevent Side Effects:

On the days you receive cyclophosphamide, you will receive mesna 4 times by vein over 15 minutes (once before, and 3 times after the cyclophosphamide infusion).

On the days you receive etoposide, you may (if needed) receive diphenhydramine by vein over 15 minutes or by mouth.

Group 3 will receive leucovorin by vein over 15 minutes, at 42 hours after the start of the methotrexate dose, and then every 6 hours until methotrexate is no longer in the body.

If your white blood cell counts become low, you may (if needed) receive filgrastim as an injection below the skin.

Study Visits:

The study visits will follow a standard schedule for tests and procedures that are done in connection with chemotherapy. At least once a week, the following tests and procedures will be performed:

* You will have a physical exam.
* Your medical history will be recorded.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.

If you are in Group 3, you will have blood drawn (about 2 teaspoons each time) for pharmacokinetic (PK) testing starting 24 hours after every methotrexate dose. This blood test will be repeated every 6 hours until the doctor decides the methotrexate level has reached a certain low level. PK testing measures the amount of study drug in the body at different time points.

Length of Study:

You may receive the study drugs for up to 6 cycles. You will be taken off the study drugs early if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

After your last dose of the study drugs:

* Blood (about 2 teaspoons) will be drawn to test your liver and kidney function.
* You will have a hearing test.
* You will have a magnetic resonance imaging (MRI) scan of the brain.

Long-Term Follow-Up:

Once you are off study, you will receive long-term follow-up from then on, according to the standard of care for brain tumors.

Other Instructions:

Before taking the study drugs, be sure to tell your doctor if:

* you have ever had any unusual or allergic reactions to any of the study drugs
* you have any type of infection (bacterial, viral, or fungal)
* you have any form of heart, kidney, liver, stomach, intestinal, or lung disease
* you have gout

For safety reasons, while you are taking the study drugs:

* Do not take any form of aspirin, ibuprofen, naproxen, or other pain relievers unless your study doctor approves.
* Do not have any alcohol (beer, wine, or liquor).
* Do not receive any vaccines unless your study doctor approves.
* Avoid contact with people who have recently taken the polio vaccine by mouth.

This is an investigational study. None of the study drugs are FDA-approved to treat choroid plexus tumors. They are all investigational for this use. Intrathecal etoposide is not FDA approved or commercially available. At this time, intrathecal etoposide is being used in research only.

Except intrathecal etoposide, all of the study drugs are FDA-approved and commercially available for use in other types of cancer:

* Etoposide by vein - for lung cancer
* Carboplatin - for ovarian cancer
* Cisplatin - for testicular cancer
* Vincristine - for leukemia
* Cyclophosphamide - for lymphoma
* Methotrexate - for leukemia
* Doxorubicin - for breast cancer
* Dactinomycin - for kidney cancer (Wilm's tumor)
* Temozolomide - for glioma (a type of brain cancer)
* Irinotecan - for colon cancer

Up to 190 patients will take part in this multicenter study. Up to 6 will be enrolled at Tufts Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of a choroid plexus tumor by a local pathologist/neuropathologist. This includes choroid plexus papilloma, atypical choroid plexus papilloma, anaplastic choroid plexus papilloma, malignant choroid plexus papilloma, and choroid plexus carcinoma.
2. Slides have been sent to the pathology reference center (by declaration of the sending center).
3. Informed consent signed
4. The first registration on the study was completed or was sent with the same mail or fax or electronic registration.
5. The reference center has confirmed the receipt of slides sent.
6. The postoperative imaging has been done and the result is available.
7. Disease status and histology: The patient is suffering from either choroid plexus carcinoma of any stage, OR an atypical choroid plexus papilloma with tumor residual after maximal possible surgical resection, OR a primary metastatic atypical choroid plexus papilloma. OR a first recurring choroid plexus papilloma that is either not resectable or was metastatic, OR a second recurrence of any choroid plexus tumor.
8. The agreement of patient or legal guardian has been documented according to the local guidelines.
9. For females in reproductive age: pregnancy test negative (both urine or blood test acceptable)
10. Females in reproductive age, patients must agree to use a medically accepted method of contraception while receiving protocol-specified medication.

Exclusion Criteria:

1. Previous chemotherapy
2. Previous radiation therapy of the central nervous system
3. White blood cell count < 2000/ uL
4. Platelet count < 85 000 / uL
5. Inadequate kidney function with Creatinine > age adapted upper normal range AND creatinine clearance or GFR determined by nuclear medicine < 70 ml/min/1.73 m2 Body surface area
6. Hearing loss more than 30 dB at 3000 Hz or more than 40 dB at 4000 Hz.
7. Echocardiography indicates myocardial dysfunction or weakness
8. Patients who are involuntarily hospitalized because of mental illness
9. Pregnancy
10. ALT or AST elevated higher than three times the upper normal level.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Wolff, MD, Principal Investigator — Pending
Locations (5):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Children's Cancer Hospital at UT MD Anderson Cancer Center, Houston, Texas
- St. Hedwig Children's Hospital, University of Regensburg (International Study Center), Regensburg, Germany
- Semmelweis University, Budapest, Hungary
- Christchurch Hospital, Christchurch, New Zealand

REFERENCES:
- See also: Neuro-Oncology 17:v186-v187, 2015. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4639153/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PI left institution prior to completion of project. 27 cases are listed in linked abstracted. (Arm A=12, Arm B=1, Arm C=4, Arm D=1, Observation = 3 and Unknown=6) PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available.
Pre-assignment Details: PI left institution prior to completion of project. 27 cases are listed in linked abstracted. (Arm A=12, Arm B=1, Arm C=4, Arm D=1, Observation = 3 and Unknown=6) PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available.
Period: Overall Study
Arm/Group | Standard Arm (1) | Doxorubicin/Cisplatin Arm (2) | Methotrexate Arm (3) | Temozolomide Irinotecan Arm (4)
Started | 12 | 1 | 4 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 12 | 1 | 4 | 1
Not completed — PI left institution, data unavailable | 12 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Population: PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available
Groups:
- Standard Arm (1): Age/Sex unknown- PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available Alternating chemotherapy cycles with etoposide 100 mg/m2 over 1 hour on days 1-5, carboplatin 350 mg/m2 over 2 hours on day 2 and 3, vincristine 1.5 mg/m2 on day 5 alternating with: etoposide 100 mg/m2 over 1 hour on days 1-5, cyclophosphamide 1 g/m2 over 1 hour on day 2 and 3, vincristine 1.5 mg/m2 on day 5. Six blocks are given in 4 week intervals (day1 to day1). Radiation is given between the second and the third cycle only to a small subgroup of patients defined by age histology staging and response to the first to cycles of chemotherapy.
- Doxorubicin/Cisplatin Arm (2): Age/Sex unknown- PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available Doxorubicin 25 mg/m²/day over 12 hrs on days 1-3, Dactinomycin 45 µg/kg/day (max. 2 mg), i.v. on day 1, and Cisplatin 70 mg/m²/d over 6 hrs on day 4, and Vincristine 1.5 mg/m²/day (max. 2 mg), i.v. on days 8, 15. An identical second cycle is started on day 28 if the side effects allow it. The further treatment is identical to the standard arm with four more cycles of chemotherapy following radiation in some of the patients in all treatment arms.
- Methotrexate Arm (3): Age/Sex unknown- PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available Methotrexate 5g/m^2 over 24 hours with leucovorin rescue at hour 42 given three times on days 1 15 and 29. The further treatment is identical in all four treatment arms.
- Temozolomide Irinotecan Arm (4): Age/Sex unknown- PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available Temozolomide is given at 150 mg/m2/day x 5 days orally and combined with irinotecan 50 mg/m2/day x 5 days as one hour infusions. Two of these cycles are followed by the common radiation - four cycle chemotherapy protocol.
- Total: Total of all reporting groups
Arm/Group | Standard Arm (1) | Doxorubicin/Cisplatin Arm (2) | Methotrexate Arm (3) | Temozolomide Irinotecan Arm (4) | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Continuous [unit: PI is no longer with the institution. Al] — PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available
Sex: Female, Male — PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: PI is no longer with the institution. All efforts have been exhausted to locate this data, but this data is no longer available
Time Frame: Till disease progression or death (up to 6 cycles of 28-day treatment)
Population: as for baseline characteristics
Arm/Group | Standard Arm (1) | Doxorubicin/Cisplatin Arm (2) | Methotrexate Arm (3) | Temozolomide Irinotecan Arm (4)
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Toxicity During First 4 Months of Therapy
Description: as for outcome 1
Time Frame: 4 Months
Population: as for baseline characteristics
Arm/Group | Standard Arm (1) | Doxorubicin/Cisplatin Arm (2) | Methotrexate Arm (3) | Temozolomide Irinotecan Arm (4)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious, and Other [Not Including Serious] Adverse Events data unavailable at sponsoring institution due to departure of PI
Description: Serious, and Other [Not Including Serious] Adverse Events data unavailable at sponsoring institution due to departure of PI
Arm/Group | Standard Arm (1) | Doxorubicin/Cisplatin Arm (2) | Methotrexate Arm (3) | Temozolomide Irinotecan Arm (4)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data unavailable at sponsoring institution due to departure of PI. Data were stored and analyzed centrally at another site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes